CLINICAL TRIAL: NCT06247410
Title: Comparative, Randomized, Open, Crossover Clinical Trial to Investigate Adhesiveness of a Newly Developed Rotigotine-containing Transdermal Patch in Patients With Parkinson's Disease
Brief Title: Clinical Trial to Investigate Patch Adhesion of Rotigotine Containing Patches in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SocraTec R&D GmbH (Other)
Collaborators: SocraMetrics GmbH (Industry); Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1402rot20ct; 2021-000867-65 (EudraCT Number)
Record Dates: First submitted 2024-01-24; First posted 2024-02-07 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Rotigotine; Rotigotine Patch; Patch Adhesion; Local Tolerability
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence: Reference-Test-Reference-Test (RTRT) (Other): Once daily patch application of one patch of Test or Reference over 4 days, i.e. a total of 4 alternating applications with RTRT sequence. Each patch remains applied for 24 h. Treatments may be directly switched without washout phase.
  Period 1: Reference: Neupro® 8 mg/24 h, 40 cm2 transdermal system containing 18 mg rotigotine (UCB Pharma GmbH, Germany), dermal application
  Period 2: Test: ROT-TDS (8 mg/24 h) 36.8 cm2 transdermal system containing 14.72 mg rotigotine (Luye Pharma AG, Germany), dermal application
  Period 3: Reference: Neupro® 8 mg/24 h, 40 cm2 transdermal system containing 18 mg rotigotine (UCB Pharma GmbH, Germany), dermal application
  Period 4: Test: ROT-TDS (8 mg/24 h) 36.8 cm2 transdermal system containing 14.72 mg rotigotine (Luye Pharma AG, Germany), dermal application
  Interventions: Drug: Rotigotine 8Mg/24Hrs Patch
- Sequence: Test-Refrence-Test-Reference (Other): Once daily patch application of one patch of Test or Reference over 4 days, i.e. a total of 4 alternating applications with TRTR sequence. Each patch remains applied for 24 h. Treatments may be directly switched without washout phase.
  Period 1: Test: ROT-TDS (8 mg/24 h) 36.8 cm2 transdermal system containing 14.72 mg rotigotine (Luye Pharma AG, Germany), dermal application
  Period 2: Reference: Neupro® 8 mg/24 h, 40 cm2 transdermal system containing 18 mg rotigotine (UCB Pharma GmbH, Germany), dermal application
  Period 3: Test: ROT-TDS (8 mg/24 h) 36.8 cm2 transdermal system containing 14.72 mg rotigotine (Luye Pharma AG, Germany), dermal application
  Period 4: Reference: Neupro® 8 mg/24 h, 40 cm2 transdermal system containing 18 mg rotigotine (UCB Pharma GmbH, Germany), dermal application
  Interventions: Drug: Rotigotine 8Mg/24Hrs Patch

INTERVENTIONS:
Drug: Rotigotine 8Mg/24Hrs Patch — Once daily patch application of one Rotigotine 8Mg/24Hrs Patch (Test or Reference) over 4 days

SUMMARY:
The investigational medicinal product (IMP) to be tested in the clinical trial (Rotigotine (ROT)-Transdermal System (TDS) (8 mg/24 h)), which is subject to this submission, was designed as a generic of Neupro® 8 mg/24 h, which is marketed in the European Union since 2006 (date of first authorisation is 2006, date of renewal of the authorisation is 2016) and serves as Reference product.

It is the intention of this clinical trial to assess patch adhesion properties of the newly developed rotigotine patch and the marketed Reference product Neupro® 8 mg/24 h after multiple patch applications.

DETAILED DESCRIPTION:
This multi-centre, open, randomized (order of treatments), multiple dose trial will be performed in a 4-period, 2-sequence-crossover design. A washout phase is not needed, i.e. the IMP application of the 2nd study period may take place the day of the IMP removal of the 1st study period (direct switch-over) and so forth.

Patients with a diagnosis of idiopathic Parkinson's disease and a continuous and stable dose of rotigotine (at least 8 mg/24 h) including use of an 8 mg/24 hours patch will be randomized.

In each of the 4 periods 1 patch, either of Test or Reference will be applied, with a release rate of 8 mg/24 h rotigotine each. Each patch will remain applied for 24 h.

Assessment of patch adhesion will be performed 5 min after application of each patch as well as at the end of the application interval prior to removal of the patch.

The clinical trial will be performed as a crossover investigation with intra-individual comparison, thus reducing variability of the patch adhesion parameters, which is supposed to be higher between patients than within an individual patient.

The patients will continue their usual medications and will only replace one 8 mg/24 h rotigotine containing patch per day with the IMPs for the duration of treatment in the clinical trial. In case of prescribed doses above 8 mg/24 h rotigotine, the remaining dose will be provided by Non-Investigational Medicinal Pproducts (NIMPs). Thus, no interruption in the prescribed dose of rotigotine will occur.

ELIGIBILITY:
Inclusion Criteria:

1. ethnic origin: Caucasian
2. age: 18 years or older
3. diagnosis of idiopathic Parkinson's disease
4. administration of a stable dose of at least 8 mg/24 h rotigotine including use of an 8 mg/24 h patch for at least 2 weeks prior to enrolment
5. agreement to refrain from swimming, bathing or using a sauna on the assessment days
6. written informed consent obtained, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the patients participating in the clinical trial

Exclusion Criteria:

Safety concerns

1. existing and/or history of significant skin hypersensitivity to adhesives or other transdermal products
2. existing and/or history of dermatitis (eczema; excluding seborrheic skin by Parkinson's disease)
3. existing and/or history of psoriasis
4. existing and/or history of an active skin disease which interferes with the rotigotine patch application according to the investigator's assessment
5. history of or current drug or alcohol dependence
6. existing medical condition or psychiatric condition which, in the opinion of the investigator, could jeopardize or compromise the patient's well-being or ability to participate in this study
7. lifetime history of suicide attempt
8. suicidal ideation in the past 6 months
9. administration of any investigational medicinal product during the last 2 months prior to individual enrolment of the patient
10. diagnosis of COVID-19 within the last 14 days prior to individual enrolment of the patient
11. contact to persons in foreign risk regions as defined by the Robert Koch Institute within the last 14 days prior to individual enrolment of the patient
12. known direct contact with insufficient protection to persons with diagnosis of COVID-19 within the last 14 days prior to individual enrolment upon reporting of the patient

    For female patients with childbearing potential only:
13. positive pregnancy test at screening examination
14. pregnant or lactating women
15. female patients who do not agree to apply highly effective contraceptive methods

    Administrative reasons
16. patients suspected or known not to follow instructions
17. patients who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Assessment of patch adhesion properties of the Test product in patients diagnosed with idiopathic Parkinson's disease at the end of the dosing interval | 24 hours
  Patch adhesion will be assessed for Test/ Reference 5 min and 23 h 55 min after patch application by trained observers. Area(s) detached will be drawn on transparent films of identical size and shape as the patch in question by the trained observer. As suggested by the Guideline on the pharmacokinetic and clinical evaluation of modified release dosage forms (EMA/CPMP/EWP/280/96 Corr1), June 2015, patch adhesion will be measured by means of the percentage of area that remains adhered at the end of the dosing interval. Additionally, the patch adhesion will be documented by taking photos at the time point of intended patch adhesion assessment of the patch and surrounding area.
  The following scores and affiliated percentages for the relative area still in tight contact with the skin will be used in order to quantify the patch adhesion:
  0 = ≥ 90% adhered
  1. = ≥ 80% adhered
  2. = ≥ 70% adhered
  3. = ≥ 60% adhered
  4. = ≥ 50% adhered
  5. = < 50% adhered or patch completely off the skin.
Comparative assessment of patch adhesion properties of the Test vs. Reference product in patients diagnosed with idiopathic Parkinson's disease at the end of the dosing interval | 24 hours
  Patch adhesion will be assessed for Test/ Reference 5 min and 23 h 55 min after patch application by trained observers. Area(s) detached will be drawn on transparent films of identical size and shape as the patch in question by the trained observer. As suggested by the Guideline on the pharmacokinetic and clinical evaluation of modified release dosage forms (EMA/CPMP/EWP/280/96 Corr1), June 2015, patch adhesion will be measured by means of the percentage of area that remains adhered at the end of the dosing interval. Additionally, the patch adhesion will be documented by taking photos at the time point of intended patch adhesion assessment of the patch and surrounding area.
  The following scores and affiliated percentages for the relative area still in tight contact with the skin will be used in order to quantify the patch adhesion:
  0 = ≥ 90% adhered
  1. = ≥ 80% adhered
  2. = ≥ 70% adhered
  3. = ≥ 60% adhered
  4. = ≥ 50% adhered
  5. = < 50% adhered or patch completely off the skin.

SECONDARY OUTCOMES:
Skin tolerability of Test and Reference based on standardised assessment of Adverse Events of Special Interest | 24 hours
  Skin irritation will be assessed for Test/ Reference 30 min after patch removal by trained observers. Skin will be visually checked and palpated. The investigator will decide based on own experience or given specifications, if a skin irritation is to be classified as Adverse Event. Additionally, photos of the skin area will be taken for documentation at all assessment time points. The following symptoms and severity grades will be used for assessment of tolerability at the site:
  Dermal response: symptom (severity); erythema (none/ minimal/ mild/ moderate/ severe); papules (none/ discrete/ pronounced); oedema (none/ minimal/ definite); vesicles (none/ non-confluent ≤ 5 mm/ confluent/ non-confluent ≥ 5 mm) Skin reaction spreading beyond site Other effects: none; slightly glazed appearance; markedly glazed appearance; glazing with peeling and cracking; glazing with fissures; film of dried serous exudates covering all or part of the site; small petechial erosions and/or scabs
Descriptive characterisation of safety and tolerability of the investigational medicinal products (IMPs) in the trial population | 4 days
  Adverse Events (AEs) observed, mentioned upon general questioning, or spontaneously reported will be documented. Adverse Events of Special Interest (AESI): Skin irritation and sensitization symptoms at patch application site Adverse Events will be listed and evaluated descriptively with regard to action taken, frequency, seriousness, intensity, relationship to the IMP, and outcome, as well as period and treatment.
  Safety parameters vital signs (BP, pulse rate (PR)): Systolic and diastolic arterial blood pressure will be measured by oscillometry using an automatic non-invasive device.
  Abnormal findings during this safety measurements, assessed as clinically relevant by the investigator, will be reported as adverse events and will be followed up and/or treated as medically appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Jost, Prof. Dr med, Principal Investigator — Parkinson-Klinik Ortenau GmbH & Co KG
Locations (8):
- Germany (8):
  - Universitätsklinikum Ulm Neur. Studienzentrale im RKU, Ulm, Baden-Wurttemberg
  - Parkinson-Klinik Ortenau GmbH & Co. KG, Wolfach, Baden-Wurttemberg
  - Neuroakademie Alzenau GbR, Alzenau in Unterfranken, Bavaria
  - Curiositas ad Sanum Studien- und Beratungs GmbH Innklinikum Haag i.OB, Haag in Oberbayern, Bavaria
  - Curiositas ad Sanum Studien- und Beratungs GmbH, München, Bavaria
  - Neurologisches Fachkrankenhaus für Bewegungsstörungen/ Parkinson, Beelitz-Heilstätten, Brandenburg
  - Gertrudis-Klinik Parkinson-Zentrum GmbH, Leun, Hesse
  - Praxis für Neurologie Dr. med. Christian Oehlwein, Gera, Thuringia

IPD SHARING:
Plan to Share IPD: No